CLINICAL TRIAL: NCT01327365
Title: Trans-Radial Percutaneous Coronary Interventions Using a Sheathless Guiding Catheter-Based Approach
Brief Title: Trans-Radial Coronary Interventions Using A Sheathless Guiding Catheter
Acronym: Sheathless-TRI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Robert F Bonvini, MD, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sheathless-TRI
Record Dates: First submitted 2010-08-23; First posted 2011-04-01 (Estimated); Last update posted 2013-03-06 (Estimated); Status verified 2013-03

CONDITIONS: Coronary Artery Disease
Keywords: significant coronary artery disease; PCI; radial approach; women; bifurcation lesion; ostial lesion; 7 Fr guiding catheter; percutaneous coronary intervention
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sheathless group (Experimental): patient randomized to the sheathless guiding catheter group
  Interventions: Procedure: trans-radial PCI (TRI)
- Conventional group (Active Comparator): patients randomized to the conventional guiding catheter group
  Interventions: Procedure: trans-radial PCI (TRI)

INTERVENTIONS:
Procedure: trans-radial PCI (TRI) — TRI performed using the sheathless guiding approach
  Arms: Sheathless group
Procedure: trans-radial PCI (TRI) — TRI performed using a conventional guiding approach
  Arms: Conventional group

SUMMARY:
Background:

The transradial approach is increasingly used in percutaneous coronary intervention (PCI) because of lower major access site complications, lower bleeding risk and earlier patient mobilization. According to this trend, in the last couple of years at the University Hospital of Geneva the investigators have changed their practice and currently the transradial approach is the most frequently used for PCI. However, the small diameter of the radial artery remains a major limitation of the technique, especially in women or for complex PCI necessitating larger bore guiding catheters. This may be overcome with sheathless guiding catheters (Asahi, Japan), allowing for a standard inner catheter diameter (6-7 Fr), with an outer diameter equivalent to a standard 5 and 6 Fr introducer sheath.

Aim:

This study is aimed to compare the transradial approach for PCI with a sheathless guiding catheter and with a standard guiding catheter in women and patients with complex lesion necessitating large bore guiding catheters.

Material and methods:

This prospective study will consecutively randomize all women and all men with bifurcation/ostial lesion of a major coronary vessel (i.e. ≈ 120/year) in whom a transradial PCI is attempted. The procedures will be performed either with a standard 6 or 7Fr guiding catheter or with the sheathless 6.5, 7.5 Fr catheters.

End-points:

Successful performance a transradial PCI in all consecutive patients which qualify according to the inclusion criteria (technical feasibility). Establish the proportion of procedures performed with no device-related complications (safety). Analyze in details the technical aspects of the sheathless catheter (efficacy).

Sample size:

The investigators have planed to include in the study ≈ 250 patients in two years. After 1 year of enrollment the investigators will perform an interim analysis and the instigators will decide at that moment, according to the observed end-points, if prolonging the study would be of any scientific value. In this case another 100 patients will be further included in the study.

Enrollment time:

The investigators will start the study as soon the local ethical committee will give us the permission. The investigators plan to start the study in July 2010. The end is expected for July 2012.

ELIGIBILITY:
Inclusion criteria:

* Patients need to be at least 18 years old.
* Patients presenting with a significant coronary artery disease who qualify for PCI and who can be treated by a radial approach.
* Any women requiring PCI who can be treated by a radial approach.
* Any patients with a bifurcation lesion or the ostial lesion of the left anterior descending (LAD) and/or left circumflex artery (LCX), lesions commonly treated with a 7 Fr guiding catheter.
* Bifurcation lesion = any lesion of a main epicardial vessel (i.e. LAD, LCX, right coronary artery) involving at least one major side branch (i.e. diagonal or marginal branches).
* Ostial lesion of the LAD or LCX = presence of a significant stenosis <5mm from the distal part of the left main.

Exclusion Criteria:

* Patients who refused to give their written informed consent.
* Male patients, in whom PCI can be easily performed with a 6 Fr standard guiding catheter (i.e. no bifurcation or ostial lesion).
* Patients in whom the radial approach is contra-indicated:

  * Patients with a dialysis arteria-venous fistula or in whom an arteria-venous fistula is planed in the future.
  * Patients with a known radial artery occlusion.
  * Patients in whom a radial approach was unsuccessfully already attempted in the past (anamnestic notion or previous medical record) secondary to a:
* Challenging vessel anatomy,
* Vessel tortuosity,
* Known impossibility to cannulate the coronary ostia by the radial approach.
* Patients in whom the Allen test results pathological bilaterally:
* In case of pathological Allen test in one hand the other hand will be tested before choosing the femoral approach.
* Patients in whom the femoral approach is adopted as primary catheterization approach (at interventionist's discretion), including:

  * Unstable patients (myocardial infarction, cardiogenic shock).
  * Patients necessitating femoral access for an intra-aortic balloon counterpulsation
  * Patients presenting with a double mammary coronary graft (right and left internal mammary utilized for by-pass grafts).
* Coronary interventions where an extreme good guiding support is mandatory (i.e. PCI of chronic total occlusion, PCI with Rotablator).
* Particularly risky PCI (e.g., PCI of the left main artery), where the femoral approach may be more comfortable for the operator.
* Patients requiring a femoral approach for a right heart catheterization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2010-08; Primary Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Procedural success | baseline
  Procedural success, defined as a successful delivery of the stent using the sheathless guding catheter, in consecutive patients according to the inclusion criteria (women and bifurcation/ostial lesions) = technical feasibility of the sheathless catheter.
Procedural safety | baseline
  Procedural safety, defined as the proportion of procedures performed in the absence of device-related complications (= safety of the sheathless catheter).
Procedural safety | +24 hours
  Procedural safety, defined as the proportion of procedures performed in the absence of device-related complications (= safety of the sheathless catheter).

SECONDARY OUTCOMES:
Safety and Tolerability | baseline
  Analyze the technical aspect of the sheathless catheter, in term of the number of Participants with Adverse Events
safety and tolerability | +24 hours
  Analyze the technical aspect of the sheathless catheter, in term of the number of Participants with Adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital, Geneva, Canton of Geneva, Switzerland

REFERENCES:
- [Background] Mamas MA, Fath-Ordoubadi F, Fraser DG. Atraumatic complex transradial intervention using large bore sheathless guide catheter. Catheter Cardiovasc Interv. 2008 Sep 1;72(3):357-364. doi: 10.1002/ccd.21637. PMID 18727126
- [Background] Mamas M, D'Souza S, Hendry C, Ali R, Iles-Smith H, Palmer K, El-Omar M, Fath-Ordoubadi F, Neyses L, Fraser DG. Use of the sheathless guide catheter during routine transradial percutaneous coronary intervention: a feasibility study. Catheter Cardiovasc Interv. 2010 Mar 1;75(4):596-602. doi: 10.1002/ccd.22246. PMID 20049959
- See also: geneva university hospital web site — http://www.hug-ge.ch